CLINICAL TRIAL: NCT04173338
Title: Phase I Study of Cabozantinib in Combination With Pemetrexed in Advanced Non-squamous Non-small Cell Lung Cancer (NSCLC), Urothelial Cancer and Advanced Malignant Mesothelioma
Brief Title: Cabozantinib With Pemetrexed in Advanced Non-small Cell Lung Cancer, Urothelial Cancer and Malignant Mesothelioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed by IRB on 3/28/22
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Nagla Abdel Karim, Professor, Hematology/Oncology, Director of Thoracic Oncology and Phase I Program, Augusta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-65
Record Dates: First submitted 2019-11-14; First posted 2019-11-21 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Non Small Cell Lung Cancer; Non-squamous Non-small-cell Lung Cancer; Urothelial Carcinoma; Malignant Mesothelioma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Transitional Cell; Mesothelioma, Malignant | interventions — cabozantinib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabozantinib + Pemetrexed (Experimental): Pemetrexed 500mg/m2 IV day 1 of each 21 day cycle + Cabozantinib 20-60mg by mouth once a day.
  Interventions: Drug: Cabozantinib; Drug: Pemetrexed

INTERVENTIONS:
Drug: Cabozantinib — start at 20mg then increase by 20mg every cycle or until there's a dose-limiting toxicity.
Drug: Pemetrexed — Start with 400mg/m2, then increase and maintain 500mg/m2 unless dose-limiting toxicity.

SUMMARY:
This study will combine cabozantinib with pemetrexed to treat patients with non-small cell lung cancer, urothelial cancer and advanced malignant mesothelioma. This study will test the safety of both drugs used together and see what effect (good or bad) it has no participants and their cancer.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced NSCLC, urothelial cancer or malignant mesothelioma.
* 18 years or older.
* At least one prior chemotherapy before entering in this trial.
* Not pregnant or breastfeeding.

Exclusion Criteria:

* Prior treatment with cabozantinib.
* Currently receiving cancer treatment (last dose 2 weeks prior to enrollment in study).
* History of bleeding disorder/bleeding history within 12 weeks before first study treatment dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Assess the maximum tolerated dose (MTD) of cabozantinib in combination with pemetrexed | 4 weeks or 28 days assessment.
  Dose-limiting toxicity of grade 3 or higher using CTCAE 5

SECONDARY OUTCOMES:
Assess objective response rate (RR) | To be measured through study completion; an average of 1 year.
  RR measured by Tumor response evaluation with RECIST
Progression-free survival (PFS) | To be measured through study completion; an average of 1 year.
  PFS measured from the time of study treatment to the date of progression.
Overall survival (OS). | OS measured through study completion, and an average of 1 year
  Measured from the time of start of treatment to time of death or time of last assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Nagla A Karim, MD, PhD, Principal Investigator — Augusta University Georgia Cancer Center
Locations (1):
- Augusta University Georgia Cancer Center, Augusta, Georgia, United States